CLINICAL TRIAL: NCT00613912
Title: Advanced MRI at 3T for the Evaluation of Ambulant Patients With Major Depression
Brief Title: Advanced MRI in Major Depression
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AUFF-2005-740-004
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Depressive Disorder, Major
Keywords: Magnetic Resonance Imaging, Magnetic Resonance Spectroscopy, Perfusion, brain
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Ambulant patients with major depression
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — * Morphological sequences
  * Arterial Spin Labelling (Perfusion)
  * Spectroscopy: anterior cingulate cortex Naa, Cho, Cr, Myo-inositol, glutamate TE 30 Reference voxel in Parietal white matter
  Other Names: 3 Tesla GE Scanner HDx

SUMMARY:
Depression is the most common psychiatric disorder.

* 3-5% of a given population has major depression.
* Less than 50% of the depressed in Denmark are diagnosed with major depression.
* 25-50% of the depressed have a relative with major depression-underlying brain pathology?

The purpose of this study is to use MRI to evaluate cerebral morphology and function in ambulant patients with major depression

DETAILED DESCRIPTION:
Previous studies within major depression, have often included hospitalized patients with severe symptoms and imaging have been performed with PET and SPECT, which uses ionizing radiation. This study focus on ambulant patients(with or without medication/ECT treatment), to find patients in an earlier stage. Cerebral perfusion with the MR sequence Arterial Spin Labelling, concentrations of different metabolites with MR spectroscopy and brain volumetry with BRAVO 3D T1 ax will be performed.

MR protocol: T2 sag, T2 FLAIR ax, ASL ax, MRS and 3D T1 ax. Scan time 45 min.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfil ICD-10´s criteria for major depression, found within the ambulant psychiatric sector and who has a HAM-D ≥ 18

Exclusion Criteria:

* If the patient has pacemaker or other magnetic devices
* Pregnancy
* Has had an operation in the brain
* bipolar disorder

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulant patients with major depression, selected from the Department of Psychatry, Aalborg hospital-Århus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Differences in morphological and functional cerebral MRI findings in patients suffering from major depression | 6 months from first MRI in each patient

CONTACTS AND LOCATIONS:
Overall Officials: Elna-Marie B Larsson, Professor, Principal Investigator — Uppsala University Hospital
Locations (1):
- Aalborg Hospital / Aarhus University Hospital, Aalborg, Jutland, Denmark